CLINICAL TRIAL: NCT05183919
Title: A Single Arm, Adaptive Design, Pivotal Trial to Assess the Efficacy of AKL-T01, a Novel Digital Intervention Designed to Improve Attention, in Adults Diagnosed With Attention Deficit Hyperactive Disorder
Brief Title: Software Treatment for Actively Reducing Severity of ADHD in Adults (STARS ADHD Adult)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Akili Interactive Labs, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Akili-057
Record Dates: First submitted 2021-12-02; First posted 2022-01-11 (Actual); Last update posted 2023-02-28 (Actual); Status verified 2023-02

CONDITIONS: Attention Deficit Hyperactivity Disorder
Keywords: ADHD
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- AKL-T01 (Experimental): Digital treatment
  Interventions: Other: Digital Treatment

INTERVENTIONS:
Other: Digital Treatment — AKL-T01 multitasking digital treatment. AKL-T01 multitasking treatment employs perceptual discrimination attention/memory task as well as a continuous motor "driving" task.

SUMMARY:
The purpose of this study is to evaluate the effects of the videogame-like digital therapy on attentional functioning and symptoms in Adults diagnosed with ADHD.

DETAILED DESCRIPTION:
This study is a multi-center, unblinded/non-controlled adaptive design study to evaluate objective attention functioning and ADHD symptoms and impairments in adults with a diagnosis of ADHD (combined or inattentive subtype), stably on or off ADHD medication, after 6 weeks of AKL-T01 treatment.

A maximum of 325 total participants from 12-30 sites will be enrolled.

During the Screening/baseline, participants will undergo screening to evaluate eligibility for the study. Eligible participants will continue onto baseline procedures in the same visit.

Treatment phase (Day 2-42) will involve using the digital therapy at home for each participant. Compliance with treatment/use requirements will be monitored remotely during this phase.

An In-Clinic assessment will be completed on Day 42 to assess key outcomes.

ELIGIBILITY:
Inclusion Criteria:

1. Adults 18 years and older
2. Diagnosis of ADHD combined or inattentive type, according to Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition (DSM-5) as confirmed by Mini International Neuropsychiatric Interview (MINI) for Attention - Deficit / Hyperactivity Disorders Studies (Adult) 7.0.2
3. Stably on or off ADHD medications for ≥4 weeks prior to study enrollment and throughout the primary 6-week study
4. Stably on or off psychoactive medications for ≥4 weeks prior to study enrollment and throughout the 6-week study
5. Baseline visit score on the ADHD-RS-IV of ≥ 24
6. Baseline visit score on the TOVA-ACS score ≤ -1.8
7. Estimated IQ score ≥80 as assessed by the Kaufmann Brief Intelligence Test, Second Edition (KBIT-II)
8. Access to and self-report of ability to connect wireless devices to a functional wireless network
9. Ability to follow written and verbal instructions (English) as assessed by the PI and/or study coordinator
10. Able to comply with all testing and study requirements
11. Completion of informed consent form

Exclusion Criteria:

1. Current controlled or uncontrolled, comorbid psychiatric diagnosis with significant symptoms that in the opinion of the Investigator may confound study data/assessments.
2. Suicidality assessed using the Columbia-Suicide Severity Rating Scale (C-SSRS)
3. Motor condition (e.g., physical deformity of the hands/arms) that prevents game playing as reported by the participant or observed by the Investigator.
4. History of moderate or severe substance use disorder within the last 12 months prior to informed consent
5. History of seizures (excluding febrile seizures), significant tics, or a current diagnosis of Tourette's Disorder.
6. Known sensitivity to playing video games, such as photo-sensitive epilepsy, light-headedness, dizziness, nausea, or motion sickness.
7. Color blindness as detected by Ishihara Color Blindness Test
8. Positive urine drug screen
9. Current or recent (3 months prior to screening) history of heavy smoking defined as the equivalent of greater than or equal to a pack of cigarettes a day
10. Any other medical condition that in the opinion of the Investigator may confound study data/assessments.
11. Participation in a clinical trial within 3 months prior to screening.
12. Previous exposure to Akili products within the 6 months prior to study enrollment
13. Plans to initiate new concomitant medications during the primary study, except for common over the counter (OTC) (e.g., ibuprofen, acetaminophen) and prescription medications (e.g., antibiotics) for minor transient ailments.
14. Planned initiation of, or significant changes in frequency, of non-pharmacological behavioral therapy during the primary study
15. Planned initiation of, or significant changes in frequency of, non-pharmacological trainings with the aim to improve cognition by means of game or app-based cognitive trainings or neurofeedback, during the primary study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 223 (Actual)
Dates: Start 2021-11-29 (Actual); Primary Completion 2023-01-13 (Actual); Study Completion 2023-01-13 (Actual)

PRIMARY OUTCOMES:
To evaluate the efficacy of AKL-T01 as determined by the change in a digitally assessed measure, Test of Variables of Attention (TOVA®) Attention Comparison Score (ACS), of sustained and selective attention, after 6 weeks of treatment with AKL-T01 | Study Day 1 to Study Day 42
  Test of Variables of Attention (TOVA)-Attention Comparison Score (ACS) of sustained and selective attention. Measures at Day 1 and Exit/Post-Treatment Visit Day 42
  TOVA ACS is a comparison of a subject's scores based on selected measures that persons with an independent diagnosis of ADHD frequently demonstrated. ACS is calculated using the following formula: TOVA ACS = Response Time Z score (Half 1) + d' Z score (Half 2) + Variability Z score (Total) + 1.80 where Response Time is the average time it takes to respond correctly to a target, d' score is a response discriminability score reflecting the ratio of hits to "false alarms", and Variability is a measure of consistency of speed of responding based on the standard deviation of the mean correct response times. A score of less than 0 indicates that the subject had similar performance to a normative ADHD population. A lower score indicates a more severe ADHD profile.

SECONDARY OUTCOMES:
To evaluate the change in ADHD symptoms, as determined by change in the ADHD Rating Scale-IV with adult prompts inattention sub-scale and total scale scores, after 6 weeks of treatment with AKL-T01 | Study Day 1 to Study Day 42
  Change in the Attention Deficit Hyperactive Disorder (ADHD) Rating Scale-IV inattention sub-scale and total scale scores. Measures taken at Baseline Visit (Day 1) and Exit/Post-Treatment Visit (Day 42).
  ADHD Rating Scale-IV is a clinician-administered questionnaire. The questionnaire is an 18-item scale that provides a rating of the severity of symptoms for Inattention and Hyperactivity-Impulsivity. The total score is obtained by adding the Inattention and Hyperactivity-Impulsivity subscale raw scores. Each item is rated on a 4-point scale; None (0), mild (1), moderate (2), severe (3). A higher score indicates more severe ADHD symptoms and behaviors.

OTHER OUTCOMES:
Change (Study Day 1 to Study Day 42) in Adult ADHD Quality of Life Questionnaire (AAQoL) total score | Study Day 1 to Study Day 42
  Change in the Adult ADHD Quality of Life Questionnaire (AAQoL) total score. Measures taken at Baseline Visit (Day 1) and Exit/Post-Treatment Visit (Day 42).
  AAQoL has 29 items to assess health-related quality of life during the past two weeks among adults with ADHD. Each item is rated by patients on a five-point Likert scale, Not at all/ Never (1) to Extremely/Very Often (5). The AAQoL has a total score and four subscale scores: Life Productivity, Psychological Health, Life Outlook, Relationships
  Total and subscale scores are computed by (1) reversing scores for all items except the seven items in the Life Outlook subscale; (2) transforming all item scores to a 0-100 point scale (1=0; 2=25; 3=50; 4=75; 5=100); and (3) summing item scores and dividing by the item count to generate subscale and total scores. The scoring algorithm indicates that the total score can be computed with up to three missing items, and each subscale score can be computed with up to one missing item.
Change (Study Day 1 to Study Day 42) in the Adult ADHD Quality of Life Questionnaire (AAQoL) Adult, subscale score for Life Productivity subscale | Study Day 1 to Study Day 42
  Change in the Adult ADHD Quality of Life Questionnaire (AAQoL) subscale score for Life Productivity. Measures taken at Baseline Visit (Day 1) and Exit/Post-Treatment Visit (Day 42).
  AAQoL has 29 items to assess health-related quality of life during the past two weeks among adults with ADHD. Each item is rated by patients on a five-point Likert scale ranging from Not at all/ Never (1) to Extremely/Very Often (5). The AAQoL has a total score and four subscale scores.
  The subscale, Life Productivity is 11 items, including getting things done on time, completing projects or tasks, remembering important things, and balancing multiple projects.
  Subscale scores are computed by (1) reversing scores for all items except the seven items in the Life Outlook subscale; (2) transforming all item scores to a 0-100 point scale (1=0; 2=25; 3=50; 4=75; 5=100); and (3) summing item scores and dividing by the item count to generate subscale scores.
Change (Study Day 1 to Study Day 42) in the Conners' Adult ADHD Rating Scales-Self Report: Short Version (CAARS-S:S) score | Study Day 1 to Study Day 42
  Change in the Conners' Adult ADHD Rating Scales-Self Report: Short Version (CAASRS:S) score. Measures taken at Baseline Visit (Day 1) and Exit/Post-Treatment Visit (Day 42).
  CAASRS:S is a Likert scale, 26-question questionnaire used to rate a patient's current functioning ability. The scores are computed by 0 = Not at all, never; 1 = Just a little, once in a while; 2 = Pretty much, often; and 3 = Very much, very frequently.
Proportion of responders at end of treatment defined as 30% reduction in total ADHD-Rating Scale-IV score | Study Day 1 to Study Day 42
  A proportion of the responders with 30% reduction in the total (ADHD) Rating Scale-IV scores. Measures taken at Baseline Visit (Day 1) and Exit/Post-Treatment Visit (Day 42).
  ADHD Rating Scale-IV is a clinician-administered questionnaire. The questionnaire is an 18-item scale that provides a rating of the severity of symptoms for Inattention and Hyperactivity-Impulsivity. The total score is obtained by adding the Inattention and Hyperactivity-Impulsivity subscale raw scores. Each item is rated on a 4-point scale; None (0), mild (1), moderate (2), severe (3). A higher score indicates more severe ADHD symptoms and behaviors.
Proportion of responders at end of treatment defined as 8-point change in Adult ADHD Quality of Life Questionnaire (AAQoL) | Study Day 1 to Study Day 42
  A proportion of the responders with an 8-point change in the Adult ADHD Quality of Life Questionnaire (AAQoL) score taken at (Day 1) and Exit/Post-Treatment Visit (Day 42).
  AAQoL has 29 items to assess health-related quality of life during the past two weeks among adults with ADHD. Each item is rated by patients on a five-point Likert scale ranging from Not at all/ Never (1) to Extremely/Very Often (5). The AAQoL yields a total score (based on all 29 items) and four subscale scores.
  Subscale scores are computed by (1) reversing scores for all items except the seven items in the Life Outlook subscale; (2) transforming all item scores to a 0-100 point scale (1=0; 2=25; 3=50; 4=75; 5=100); and (3) summing item scores and dividing by the item count to generate subscale and total scores. The scoring algorithm indicates that the total score can be computed with up to three missing items, and each subscale score can be computed with up to one missing item.
Change (Study Day 1 to Study Day 42) in TOVA metrics other than ACS, Ex-Gaussian Tau Total | Study Day 1 to Study Day 42
  To evaluate changes in the following additional Test of Variables of Attention (TOVA) metrics other than Attention Comparison Score (ACS) - Ex-Gaussian Tau.
  TOVA is a comparison of a subject's scores based on selected measures that persons with an independent diagnosis of ADHD frequently demonstrated.
  TOVA metric evaluated for change is:
  Ex-Gaussian Tau: The exponential decay (or "right hand tail") of the correct response times, modeled using the Ex-Gaussian distribution. Total refers to entire test (both H1 and H2). H1 refers to the first half of the test where target stimulus is infrequent (1 target to 3.5 non-targets), and H2 represents the second half where target stimulus is frequent (3.5 targets to 1 non-target).
  Measures at Day 1 and Exit/Post-Treatment Visit Day 42.
Change (Study Day 1 to Study Day 42) in TOVA metrics other than ACS, Commission Errors Standard Score H2 | Study Day 1 to Study Day 42
  To evaluate changes in the following additional Test of Variables of Attention (TOVA) metrics other than Attention Comparison Score (ACS) - Commission Errors Standard.
  TOVA is a comparison of a subject's scores based on selected measures that persons with an independent diagnosis of ADHD frequently demonstrated.
  TOVA metric evaluated for change is:
  Commission Errors Standard Score H2: Commission errors are the number of times the patient clicked the microswitch at the incorrect time. H2 represents the second half where target stimulus is frequent (3.5 targets to 1 non-target).
  Measures at Day 1 and Exit/Post-Treatment Visit Day 42.
Change (Study Day 1 to Study Day 42) in TOVA metrics other than ACS, Response Time Variability Standard Score Total | Study Day 1 to Study Day 42
  To evaluate changes in the following additional Test of Variables of Attention (TOVA) metrics other than Attention Comparison Score (ACS) - Response Time Variability Standard Score Total.
  TOVA is a comparison of a subject's scores based on selected measures that persons with an independent diagnosis of ADHD frequently demonstrated.
  TOVA metric evaluated for change is:
  Response Time Variability Standard Score Total: The standard score for the first standard deviation of the correct response times. Total refers to entire test (both H1 and H2). H1 refers to the first half of the test where target stimulus is infrequent (1 target to 3.5 non-targets), and H2 represents the second half where target stimulus is frequent (3.5 targets to 1 non-target).
  Measures at Day 1 and Exit/Post-Treatment Visit Day 42.
Change (Study Day 1 to Study Day 42) in TOVA metrics other than ACS, Response Time Mean Standard Score H1 | Study Day 1 to Study Day 42
  To evaluate changes in the following additional Test of Variables of Attention (TOVA) metrics other than Attention Comparison Score (ACS) - Response Time Mean Standard Score H1.
  TOVA is a comparison of a subject's scores based on selected measures that persons with an independent diagnosis of ADHD frequently demonstrated.
  TOVA metric evaluated for change is:
  Response Time Mean Standard Score H1:The standard score for the mean response time of the correct responses. H1 refers to the first half of the test where target stimulus is infrequent (1 target to 3.5 non-targets).
  Measures at Day 1 and Exit/Post-Treatment Visit Day 42.
Change (Study Day 1 to Study Day 42) in TOVA metrics other than ACS, D-Prime Standard Score H2 | Study Day 1 to Study Day 42
  To evaluate changes in the following additional Test of Variables of Attention (TOVA) metrics other than Attention Comparison Score (ACS) - D-Prime Standard Score H2.
  TOVA is a comparison of a subject's scores based on selected measures that persons with an independent diagnosis of ADHD frequently demonstrated.
  TOVA metric evaluated for change is:
  D-Prime Standard Score H2: D-Prime score is a response discriminability score reflecting the ratio of hits to false alarms. The measure is derived from Signal Detection Theory and has been shown to help distinguish non-impaired individuals from those diagnosed with attention disorders. The score reflects the accuracy of target (signal) and nontarget (noise) discrimination and can be interpreted as a measure of perceptual sensitivity. H2 represents the second half where target stimulus is frequent (3.5 targets to 1 non-target).
  Measures at Day 1 and Exit/Post-Treatment Visit Day 42.
Change (Study Day 1 to Study Day 42) in TOVA metrics other than ACS, Omission Errors Standard Score H2 | Study Day 1 to Study Day 42
  To evaluate changes in the following additional Test of Variables of Attention (TOVA) metrics other than Attention Comparison Score (ACS) - Omission Errors Standard Score H2.
  TOVA is a comparison of a subject's scores based on selected measures that persons with an independent diagnosis of ADHD frequently demonstrated.
  TOVA metric evaluated for change is:
  Omission Errors Standard Score H2: Omission Errors are the number of times the patient failed to click the microswitch when the target was presented. H2 represents the second half where target stimulus is frequent (3.5 targets to 1 non-target).
  Measures at Day 1 and Exit/Post-Treatment Visit Day 42.

CONTACTS AND LOCATIONS:
Locations (14):
- United States (14):
  - Melmed Center, Scottsdale, Arizona
  - CNS Clinical Research Trials, Garden Grove, California
  - Innovative Clinical Research, Inc., Lauderhill, Florida
  - Accel Research Sites, Maitland, Florida
  - Behavioral Clinical Research, Inc., Miami Lakes, Florida
  - Midwest Research Group, Saint Charles, Missouri
  - Alivation Research, Lincoln, Nebraska
  - Center for Psychiatry and Behavioral Medicine, Inc., Las Vegas, Nevada
  - Hassman Research Institute, Berlin, New Jersey
  - Albuquerque Neuroscience, Inc., Albuquerque, New Mexico
  - MindPath Care Centers, Raleigh, North Carolina
  - IPS Research, Oklahoma City, Oklahoma
  - FutureSearch Trials, Dallas, Texas
  - Southeast Houston Research, Inc., Houston, Texas

REFERENCES:
- [Derived] Stamatis CA, Heusser AC, Simon TJ, Ala'ilima T, Kollins SH. Real-time cognitive performance metrics derived from a digital therapeutic for inattention predict ADHD-related clinical outcomes: Replication across three independent trials of AKL-T01. Transl Psychiatry. 2024 Aug 11;14(1):328. doi: 10.1038/s41398-024-03045-0. PMID 39128918
- [Derived] Flannery JE, Hinshaw SP, Kollins SH, Stamatis CA. Secondary analyses of sex differences in attention improvements across three clinical trials of a digital therapeutic in children, adolescents, and adults with ADHD. BMC Public Health. 2024 Apr 29;24(1):1195. doi: 10.1186/s12889-024-18597-5. PMID 38685016